CLINICAL TRIAL: NCT02793817
Title: A Phase 3, Double-Masked, Randomized, Controlled Study to Evaluate the Safety and Efficacy of KPI-121 1.0% Ophthalmic Suspension in Subjects With Postsurgical Inflammation and Pain
Brief Title: Safety and Efficacy of KPI-121 in Subjects With Postsurgical Inflammation and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-005
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2018-10

CONDITIONS: Post Surgical Ocular Inflammation and Pain
Keywords: postsurgical; postoperative; ocular; cataract; inflammation; pain; corticosteroid
MeSH Terms: conditions — Pain; Cataract; Inflammation | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KPI-121 1.0% Ophthalmic Suspension (Active Comparator): dosed BID
  Interventions: Drug: KPI-121 1% Ophthalmic Suspension dosed BID
- Vehicle of KPI-121 Ophthalmic Suspension (Placebo Comparator): dosed BID
  Interventions: Drug: Vehicle of KPI-121 Ophthalmic Suspension dosed BID

INTERVENTIONS:
Drug: KPI-121 1% Ophthalmic Suspension dosed BID
  Other Names: Loteprednol etabonate
  Arms: KPI-121 1.0% Ophthalmic Suspension
Drug: Vehicle of KPI-121 Ophthalmic Suspension dosed BID
  Other Names: Placebo
  Arms: Vehicle of KPI-121 Ophthalmic Suspension

SUMMARY:
The primary objective of the study is to investigate the efficacy and safety of KPI-121 1.0% ophthalmic suspension compared to placebo in subjects who have undergone cataract surgery.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, double-masked, randomized, placebo-controlled, parallel-group study designed to evaluate the efficacy and safety of KPI-121 1.0% ophthalmic suspension versus placebo in subjects who require treatment of postoperative anterior ocular inflammation.

ELIGIBILITY:
Inclusion Criteria:

Candidates for routine, uncomplicated cataract surgery

In Investigator's opinion, potential postoperative Snellen Distance VA by pinhole method of at least 20/200 in study eye.

Exclusion Criteria:

* Known hypersensitivity/contraindication to study product(s) or components.
* History of glaucoma, intraocular pressure (IOP) >21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; severe/serious systemic disease or uncontrolled medical condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within the 30 days prior to screening or 18 days following surgery.
* In the opinion of Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Arizona Eye Center, Chandler, Arizona
  - Cornea and Cataract Consultants of CA, Phoenix, Arizona
  - Sall Research Medical Center, Artesia, California
  - Orange County Ophthalmology, Garden Grove, California
  - Lugene Eye Institute, Glendale, California
  - Inland Eye Specialists, Hemet, California
  - United Medical Research Institute, Inglewood, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Pendleton Eye Center, Oceanside, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Arch Health Partners, Poway, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc, Redding, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Shettle Eye Research, Inc, Largo, Florida
  - International Research Center, Tampa, Florida
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Jacksoneye, S. C., Lake Villa, Illinois
  - The Eye Care Institute, Louisville, Kentucky
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - Comprehensive Eye Care, Ltd. / Vision Research Institute, LLC, Washington, Missouri
  - Abrams Eye Institute, Las Vegas, Nevada
  - Duke University Eye Center, Durham, North Carolina
  - Apex Eye, Cincinnati, Ohio
  - Roseburg Research Associates, LLC, Roseburg, Oregon
  - Eye Care Specialists, Kingston, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina
  - Texan Eye, PA / Keystone Research, Ltd, Austin, Texas
  - The Cataract & Glaucoma Center, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Kozlovsky Delay & Winter Eye Consultants, LLC Corona Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KPI-121 1.0% Ophthalmic Suspension: dosed BID
  KPI-121 1% Ophthalmic Suspension dosed BID
- Vehicle of KPI-121 Ophthalmic Suspension: dosed BID
  Vehicle of KPI-121 Ophthalmic Suspension dosed BID
Period: Overall Study
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | Vehicle of KPI-121 Ophthalmic Suspension
Started | 261 | 259
Completed | 258 | 254
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | Vehicle of KPI-121 Ophthalmic Suspension | Total
Number analyzed (Participants) | 261 | 259 | 520
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [38 to 89] | 69.3 [40 to 90] | 68.4 [38 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 144 | 288
  Male | 117 | 115 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 36 | 74
  Not Hispanic or Latino | 223 | 223 | 446
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 27 | 24 | 51
  White | 206 | 207 | 413
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 261 | 259 | 520

OUTCOME MEASURES:

1. Primary Outcome: Complete Resolution of Anterior Chamber (AC) Cells at Day 8
Description: Number and percentage of subjects with complete resolution of AC cells in the surgical eye (study eye) at Day 8 maintained through Day 15, without receiving rescue medication prior to Day 15, for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. = 1 - 5 cells
  2. = 6 - 15 cells
  3. = 16 - 30 cells
  4. = greater than 30 cells
Time Frame: Visit 5 (Day 8) maintained through Visit 6 (Day 15)
Population: Intent to Treat - All subjects randomized
Measure: Count of Participants; unit: Participants
Groups:
- KPI-121 1% Ophthalmic Suspension: KPI-121 1% Ophthalmic Suspension dosed BID
- Vehicle of KPI-121 1% Ophthalmic Suspension: Vehicle of KPI-121 1% Ophthalmic Suspension dosed BID
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 261 | 259
Participants | 54 | 32
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; P-values were based on 2-sided chi-squared tests (unadjusted) wherein the a priori significance level was 0.05; Test type: Superiority; p = 0.0105, Chi-squared — To account for multiplicity, a step-down testing procedure was applied, whereby inference for a test in the pre-defined hierarchy was dependent upon statistical significance having been demonstrated for the previous test in the hierarchy; Without adjustment for any covariates; Difference in percentage of responders = 8.3, 95% CI 2-sided [2.0 to 14.7] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

2. Primary Outcome: Complete Resolution of Ocular Pain at Day 8
Description: Number and percentage of subjects with complete resolution of ocular pain in the surgical eye (study eye) at Day 8 maintained through Day 15, without receiving rescue medication prior to Day 15, for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Subjects were given the Subject-Rated Ocular Pain Assessment to subjectively rate their pain at Days 1, 4, 8, 15, and the follow-up visit between Days 17 and 19. Higher scores were worse outcomes.
  The following scoring scale was used for ocular pain:
  0 = None
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Moderately Severe
  5. = Severe
Time Frame: Visit 5 (Day 8) maintained through Visit 6 (Day 15)
Population: Intent to Treat - All subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 261 | 259
Participants | 149 | 96
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; P-values were based on 2-sided chi-squared test (unadjusted), wherein a priori significance level was 0.05; Test type: Superiority; p < 0.0001, Chi-squared — To account for multiplicity, a step-down closed testing procedure was applied, whereby inference for a test in the pre-defined hierarchy was dependent upon statistical significance having been demonstrated for the previous test in the hierarchy; Without adjustment for any covariates; Difference in percentage of responders = 20.0, 95% CI 2-sided [11.6 to 28.4] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

3. Secondary Outcome: Complete Resolution of Ocular Pain at Day 4
Description: Number and percentage of subjects with complete resolution of ocular pain in the surgical eye (study eye) at Day 4 maintained through Day 15, without receiving rescue medication prior to Day 15, for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Subjects were given the Subject-Rated Ocular Pain Assessment to subjectively rate their pain at Days 1, 4, 8, 15, and the follow-up visit between Days 17 and 19. Higher scores were worse outcomes.
  The following scoring scale was used for ocular pain:
  0 = None
  1. = Minimal
  2. = Mild
  3. = Moderate
  4. = Moderately Severe
  5. = Severe
Time Frame: Visit 4 (Day 4) maintained through Visit 6 (Day 15)
Population: Intent to Treat - All subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 261 | 259
Participants | 109 | 64
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; Test type: Superiority; p < 0.0001, Chi-squared — P-value was based on a 2-sided chi-squared test (unadjusted) wherein the a priori significance level was 0.0167 for each secondary endpoint. Overall alpha for all secondary endpoints was controlled at 0.05; Without adjustment for any covariates; Difference in percentage of responders = 17.1, 95% CI 2-sided [9.1 to 25.0] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

4. Secondary Outcome: Complete Resolution of Anterior Chamber (AC) Flare at Day 4
Description: Number and percentage of subjects with complete resolution of AC flare in the surgical eye (study eye) at Day 4 maintained through Day 15, without receiving rescue medication prior to Day 15, for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Investigators were asked to grade AC flare based on the following scale wherein higher scores indicate a higher degree of flare present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Flare 0 = None
  1. = Mild (trace to clearly noticeable, visible)
  2. = Moderate (without plastic aqueous humor)
  3. = Marked (with plastic aqueous humor)
  4. = Severe (with fibrin deposits and/or clots)
Time Frame: Visit 4 (Day 4) maintained through Visit 6 (Day 15)
Population: Intent to Treat - All subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 261 | 259
Participants | 113 | 63
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 3, analysis 1]; Without adjustment for any covariates; Difference in percentage of responders = 19.0, 95% CI 2-sided [11.0 to 26.9] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

5. Secondary Outcome: Change From Baseline (BL) Anterior Chamber (AC) Cells at Day 4
Description: The difference in mean changes from BL in AC cell count grade at Day 4 for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. = 1 - 5 cells
  2. = 6 - 15 cells
  3. = 16 - 30 cells
  4. = greater than 30 cells
Time Frame: Visit 1 (Baseline) and Visit 4 (Day 4)
Population: Intent to Treat - All subjects randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 258 | 257
score on a scale | -0.7 (0.84) | -0.5 (0.91)
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; P-value was based on a 2-sided chi-squared test (unadjusted) wherein the a priori significance level was 0.0167 for each secondary endpoint. Overall alpha for all secondary endpoints was controlled at 0.05; Test type: Superiority; p = 0.0078, Chi-squared; Without adjustment for any covariates; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.31 to -0.05] — Estimated Value is the between-group difference for change from BL

6. Post Hoc Outcome: Change From Baseline (BL) Anterior Chamber (AC) Cells at Day 8
Description: The difference in mean changes from BL in AC cell count grade at Day 8 for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. = 1 - 5 cells
  2. = 6 - 15 cells
  3. = 16 - 30 cells
  4. = greater than 30 cells
Time Frame: Visit 1 (Baseline) and Visit 5 (Day 8)
Population: Intent to Treat - All subjects randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 258 | 257
score on a scale | -1.3 (0.90) | -1.0 (0.94)
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; Test type: Superiority; p = 0.0005, Chi-squared — P-values have no inferential value for post hoc evaluations; Without any adjustment for covariates; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.38 to -0.11] — Estimated Value is the between-group difference in change from BL

7. Post Hoc Outcome: Change From Baseline (BL) Anterior Chamber (AC) Cells at Day 15
Description: The difference in mean changes from BL in AC cell count grade at Day 15 for KPI-121 1% dosed twice daily (BID) compared with vehicle dosed BID.
  Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. = 1 - 5 cells
  2. = 6 - 15 cells
  3. = 16 - 30 cells
  4. = greater than 30 cells
Time Frame: Visit 1 (Baseline) and Visit 6 (Day 15)
Population: Intent to Treat - All subjects randomized
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
Number analyzed (Participants) | 257 | 254
score on a scale | -1.8 (0.84) | -1.6 (0.87)
Statistical Analysis 1: Comparison: KPI-121 1% Ophthalmic Suspension vs Vehicle of KPI-121 1% Ophthalmic Suspension; Test type: Superiority; p = 0.0169, Chi-squared — P-values have no inferential value for post hoc evaluations; Without adjustments for any covariates; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.28 to -0.03] — Estimated Value is the between-group difference for change from BL

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a subjects signed the informed consent until they exited the study at the end of Visit 7 (up to 18 days).
Arm/Group | KPI-121 1% Ophthalmic Suspension | Vehicle of KPI-121 1% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/259
Serious Adverse Events (participants affected / at risk) | 1/261 | 2/259
Other Adverse Events (participants affected / at risk) | 18/261 | 21/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 1% Ophthalmic Suspension (N=261) | Vehicle of KPI-121 1% Ophthalmic Suspension (N=259)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
erebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 1% Ophthalmic Suspension (N=261) | Vehicle of KPI-121 1% Ophthalmic Suspension (N=259)
Cystoid macular oedema (Eye disorders) | 3 (3) | 3 (4)
Eye pain (Eye disorders) | 3 (3) | 6 (6)
Posterior capsule opacification (Eye disorders) | 3 (3) | 4 (4)
Instilation site pain (General disorders) | 1 (2) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No submission for publication or public disclosure will be made by the PI until after the publication of the results of the multi-center clinical trial by the Sponsor. Thereafter, PI shall provide KALA with an advance copy of any proposed publication or public disclosure at least sixty (60) days prior to the planned date of submission or disclosure and KALA shall have forty-five (45) days from the date of its receipt to recommend changes.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02793817/Prot_SAP_002.pdf